CLINICAL TRIAL: NCT01944514
Title: Improving Risk Stratification of Patients for Implantable Cardioverter Defibrillators Through Electrophysiological Tests, Cardiac Magnetic Resonance Imaging, Autonomic Function Tests, RNA Analysis and Plasma Biomarkers.
Brief Title: Implantable Cardioverter Defibrillators - Improving Risk Stratification
Acronym: ICD-IRS
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: University of Leicester (Other); Da Vinci Health Technology Innovation Network (Other); LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: UHL-10824: ICD-IRS
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Sudden Cardiac Death; Implantable Defibrillator User; Myocardial Infarction; Arrhythmias, Cardiac
Keywords: Action potential duration restitution; Ventricular arrhythmia; Sudden cardiac death; Peri-infarct zone; Electrocardiogram
MeSH Terms: conditions — Death, Sudden, Cardiac; Myocardial Infarction; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh frozen plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ischaemic cardiomyopathy group: Patients with ischaemic cardiomyopathy attending for ICD implantation / Ventricular tachycardia stimulation testing as part of ICD risk stratification
- Non-ischaemic cohort: Patients attending for ICD implantation / ventricular tachycardia stimulation test who do not have ischaemic cardiomyopathy.
- Control group: Patients attending for electrophysiological study with no conditions that place them at risk of sudden cardiac death.

SUMMARY:
Worldwide three million people a year die from sudden cardiac death (SCD). In most cases there is no warning and the heart is stopped by a sudden arrhythmia. We know that some people are at high risk of sudden cardiac death and can prevent their deaths with an implantable cardioverter defibrillator (ICD) that is implanted in a minor operation.

However, most people who die from sudden cardiac death are not found to be at high risk by our current risk markers and 40% of the people who have ICDs do not have therapy within the first 4 years after implant. We need new and better ways of identifying people who are at high risk of sudden cardiac death so that we can prevent their deaths with ICDs. Our understanding of the electrical signals in the heart has increased considerably in recent years; in no small part this is due to our Principal Investigator Professor Andre Ng's basic science work. This study aims to take the understanding of action potential duration (APD) restitution gained through our work and other studies in humans and in computer simulations and translate it into a fresh way of assessing risk of sudden cardiac death.

This study will carefully examine electrical activity, using APD restitution, in the hearts of patients who are having ICDs fitted because of their high risk of sudden cardiac death and combine this with a detailed heart scan, assessment of autonomic nervous system and gene expression data. We will then follow these patients up to see who benefits from their ICD. This wide ranging information will give us as complete a picture as possible of the factors that cause sudden cardiac death. We hope to use this to identify better predictors of sudden cardiac death.

The study hypotheses are as follows:

Primary

1. Regional Restitution Instability Index (R2I2) will be significantly higher in patients reaching the endpoint of ventricular endpoint / sudden cardiac death than in those not.
2. An R2I2 cut-off of 1.03 will partition patients into high and low risk groups.

   Secondary
3. Peri-infarct zone mass in grams will be significantly higher in patients reaching the endpoint of ventricular endpoint / sudden cardiac death than in those not.

ELIGIBILITY:
Inclusion Criteria:

* Attending for ICD implantation under NICE criteria or attending for an ICD box-change procedure or attending for an Electrophysiological test as part of NICE assessment for ICD implantation
* Age >18
* History of ischaemic heart disease or non-ischaemic cardiomyopathy or inherited sudden cardiac death syndrome.

Exclusion Criteria:

* <28 days since acute coronary syndrome / cardiac surgery
* Unable to give informed consent
* Women who are pregnant / planning pregnancy
* Contraindication for defibrillator safety margin test

  * Haemodynamic instability
  * Severe valvular heart disease
  * Symptomatic, severe, coronary artery disease
  * Recent stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ischaemic cardiomyopathy cohort: patients with a history of myocardial infarction attending for ICD implantation / Ventricular tachycardia stimulation test.
  Non-Ischaemic cohort: patients without a history of myocardial infarction attending for ICD implantation / Ventricular tachycardia stimulation test.
  Control group: Patients with normal hearts and no conditions / family history that increases risk of sudden cardiac death attending for an electrophysiological study.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Regional Restitution Instability Index | 18months - 2years
  Regional Restitution Instability Index (R2I2) is a measure of electrical instability. R2I2 is calculated as the mean of the standard deviation of the residuals from the mean gradients for each ECG lead across a range of diastolic intervals. An R2I2 cut-off of 1.03 (no units) will partition the study population into high and low risk groups.

SECONDARY OUTCOMES:
Peri-infarct zone | 18months-2 years
  Peri-infarct zone is calculated from cardiac magnetic resonance imaging scans with late gadolinium enhancement. The full width half maximum technique will be used and Peri-infarct zone assessed using peri-infarct zone mass in grams.

CONTACTS AND LOCATIONS:
Overall Officials: G. Andre Ng, MBCHb, PhD, Principal Investigator — University of Leicester

REFERENCES:
- [Background] Nicolson WB, McCann GP, Brown PD, Sandilands AJ, Stafford PJ, Schlindwein FS, Samani NJ, Ng GA. A novel surface electrocardiogram-based marker of ventricular arrhythmia risk in patients with ischemic cardiomyopathy. J Am Heart Assoc. 2012 Aug;1(4):e001552. doi: 10.1161/JAHA.112.001552. Epub 2012 Aug 24. PMID 23130163
- [Derived] Nicolson WB, McCann GP, Smith MI, Sandilands AJ, Stafford PJ, Schlindwein FS, Samani NJ, Ng GA. Prospective evaluation of two novel ECG-based restitution biomarkers for prediction of sudden cardiac death risk in ischaemic cardiomyopathy. Heart. 2014 Dec;100(23):1878-85. doi: 10.1136/heartjnl-2014-305672. Epub 2014 Aug 4. PMID 25092878